CLINICAL TRIAL: NCT00363116
Title: An Open-Label, Comparative Trial of Two Daclizumab Dosing Strategies Versus No Induction Treatment in Combination With Tacrolimus, Mycophenolate Mofetil, and Steroids for the Prevention of Acute Allograft Rejection in Simultaneous Kidney/Pancreas Transplant Recipients
Brief Title: A Trial of Two Daclizumab Dosing Strategies vs. No Induction Treatment With Tacrolimus, Mycophenolate Mofetil , & Steroids for the Prevention of Acute Allograft Rejection in Simultaneous Kidney/Pancreas Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Roche Pharma AG (Industry); University of Tennessee (Other)
Responsible Party: Principal Investigator, Rita Alloway, Investigator, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZEN049
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Acute Allograft Rejection in Simultaneous Kidney/Pancreas Transplant Recipients
Keywords: Kidney transplant; Pancreas transplant; Daclizumab; Tacrolimus; Mycophenolate mofetil; Steroids; Immunosuppression; Acute allograft rejection
MeSH Terms: interventions — Daclizumab

ARMS (3):
- 5 Dose Daclizbumab (Active Comparator): daclizumab 1 mg/kg/dose every 14 days for 5 doses
  Interventions: Drug: Daclizumab
- 2 Dose Daclizaumab (Active Comparator): daclizumab 2 mg/kg/dose every 14 days for 2 doses
  Interventions: Drug: Daclizumab
- Control (Active Comparator): no antibody induction
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Daclizumab — daclizumab 1 mg/kg/dose every 14 days for 5 doses

SUMMARY:
The purpose of the study is to determine the safety and efficacy of two dosing regimens of daclizumab in simultaneous kidney/pancreas transplant recipients.

DETAILED DESCRIPTION:
The purpose of the study is to determine the safety and efficacy of two dosing regimens of daclizumab as an adjunctive immunosuppressive agent in simultaneous kidney/pancreas transplant recipients receiving tacrolimus, mycophenolate mofetil, and steroids as primary maintenance immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Simultaneous kidney/pancreas transplant recipients
* Insulin dependent Type 1 or 2 diabetes pretransplant
* Recipient age 18-65 years
* Donor age 5-65 years
* Women must have negative serum pregnancy test and practice birth control for study duration
* Negative T-cell crossmatch
* Parent (or guardian) is able to understand the consent form and give written informed consent

Exclusion Criteria:

* Prior treatment with daclizumab
* Known sensitivity or contraindication to tacrolimus, MMF, or steroids
* Patient with significant or active infection
* Patients with a positive lymphocytotoxic crossmatch using donor lymphocytes and recipient serum
* Patients whose life expectancy is severely limited by diseases other than renal disease
* Ongoing substance abuse, drug or alcohol
* Major ongoing psychiatric illness or recent history of noncompliance
* Insufficient cardiovascular reserve
* Malignancy within last 5 years, excluding nonmelanoma skin cancers
* Serologic evidence of infection with HIV or Hepatitis B surface antigen positive
* Investigational drug within 30 days prior to transplant surgery
* Anti-T cell therapy within 30 days prior to transplant surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 1999-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of presumed acute kidney or pancreas rejection, death, and kidney or pancreas graft loss in the first 6 months post transplant.

SECONDARY OUTCOMES:
Incidence, timing and severity of fungal infections.
Incidence, timing and severity of malignancies.
Hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Stratta, MD, Principal Investigator — University of Tennessee
Locations (24):
- United States (23):
  - University of California - Davis, Davis, California
  - University of California - Los Angeles, Los Angeles, California
  - Washington Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, College Park, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Cornell University, Ithaca, New York
  - Carolina Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - University of Texas - Houston, Houston, Texas
  - Baylor University, Waco, Texas
  - Medical College of Virginia, Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Toronto Hospital, Toronto, Ontario, Canada